CLINICAL TRIAL: NCT05201443
Title: Clinical and Biochemical Evaluation of the Efficacy of Non-Surgical Treatment Approaches in the Treatment of Peri-implantitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nazan Ece Erduran, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-19059
Record Dates: First submitted 2021-10-12; First posted 2022-01-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diode Laser (Experimental): At baseline, diode laser is applied to one group.
  Interventions: Device: Diode laser; Device: Titanium curettes
- Titanium curettes (Active Comparator): At baseline, titanium curettes are used to both of the groups
  Interventions: Device: Titanium curettes

INTERVENTIONS:
Device: Diode laser — Diode Laser is applied to one group as an adjunctive therapy.
  Arms: Diode Laser
Device: Titanium curettes — Non-surgical treatment with titanium curettes were administrated to both groups.

SUMMARY:
Peri-implantitis is a pathological condition associated with plaque that develops around dental implants, characterized by inflammation and progressive bone loss in the peri-implant area. Bleeding on probing, suppuration, increased pathological pocket depths and/or mucosal recessions are seen with radiographic bone loss in peri-implantitis. When evaluated histologically, the lesion extends to the apical part of the pocket epithelium and contains a large amount of plasma cells, macrophages and neutrophils. In the Peri-implant crevicular fluid analysis, which is one of the most important parameters that enable the biochemical and immunological evaluation of the inflammatory state in the peri-implant region, information about the current inflammatory situation can be obtained by evaluating the content of an osmotic inflammatory exudate originating from the vessels in the gingival plexus. Many surgical and non-surgical methods have been proposed for the treatment of peri-implantitis. Mechanical surface debridement, laser application and air abrasives are a part of non-surgical treatment of peri-implantitis. In this study, we examined the effectiveness of diode laser in addition to mechanical debridement with titanium curettes. In our study, we aimed to compare these two treatments biochemically by determining the changes in interleukin-1β, Interleukin-10, Interleukin-17, RANKL, osteoprotegerin, TWEAK and sclerostin biomarkers in Peri-implant crevicular fluid and clinically.

DETAILED DESCRIPTION:
Primary outcome measures (probing depth as clinical parameter) and secondary outcome measures ( collection of gingival crevicular fluid, gingival bleeding time index, gingival index, plaque index and clinical attachment level) asre recorded in baseline, third and sixth month. The change between these parameters is observed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 5mm or more peri-implant pockets
* Not having periodontal treatment in the last 3 months,
* The informed consent form must be approved,
* At least 18 years old.

Exclusion Criteria:

* Presence of systemic disease,
* Smoking,
* Regular use of non-steroidal anti inflammatory drugs,
* Having been treated with antibiotics in the last 3 months,
* Individuals in need of pre-treatment antibiotic prophylaxis,
* Pregnancy and lactation,
* Not approving the informed consent form,
* Patients with known allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Clinical parameter probing depth | Baseline, 3 months and 6 months
  The primary outcome of the study was the control examination performed 3 months after the first examination. Probing depth was measured with a periodontal probe by the distance between gingival margin and the base of the pocket. The change between these time frames are recorded.

SECONDARY OUTCOMES:
Another outcome of the study is the collection of gingival crevicular fluid samples in the 3rd month. | Baseline, 3 months and 6 months
  Samples are obtained by means of paper strips placed gently in the gingival groove. These samples are stored at -20 ° C for later analysis by ELISA method. The change between these time frames are recorded.
Gingival bleeding time index | Baseline, 3 months and 6 months
  Bleeding on probing according to the time is recorded. The change between these time frames are recorded.
Gingival index | Baseline, 3 months and 6 months
  The gingival index is graded as follows:
  0 = Normal gingiva
  1. Mild inflammation, slight change in color, slight oedema. No bleeding on probing
  2. Moderate inflammation redness, oedema and glazing. Bleeding on probing
  3. Severe inflammation marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
Plaque index | Baseline, 3 months and 6 months
  0 = No plaque in the gingival area.
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Clinical attachment level | Baseline, 3 months and 6 months
  The distance in millimeters from the cemento-enamel junction to the bottom of the pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Güliz Nigar GÜNCÜ, Prof. Dr., Study Director — study director; Abdullah Cevdet AKMAN, Prof Dr, Principal Investigator — Principal Investigator; Rahime Meral NOHUTCU, Principal Investigator — Principal Investigator; Ali Tuğrul GÜR, Phd, Principal Investigator — Principal Investigator; Aslı PINAR, Prof Dr, Principal Investigator — biochemistry
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)